CLINICAL TRIAL: NCT07060664
Title: Review of Proximal Humerus Fracture Outcomes
Brief Title: Study on Outcomes of Proximal Humerus Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Gregory Iovanel, Principal Investigator, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00002567
Record Dates: First submitted 2025-06-29; First posted 2025-07-11 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Proximal Humerus Fracture
Keywords: proximal humerus fracture; humerus; fracture; shoulder; ORIF; IMN; nail; open reduction internal fixation
MeSH Terms: conditions — Fractures, Bone | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative Management (Active Comparator)
  Interventions: Procedure: open reduction internal fixation; Procedure: intramedullary nail; Procedure: reverse total shoulder arthroplasty
- Non-operative Management (No Intervention)

INTERVENTIONS:
Procedure: open reduction internal fixation — treatment with open reduction and plates/screws
  Other Names: ORIF
  Arms: Operative Management
Procedure: intramedullary nail — open reduction and intramedullary nail
  Other Names: IMN
  Arms: Operative Management
Procedure: reverse total shoulder arthroplasty — reverse total shoulder arthroplasty
  Other Names: RTSA
  Arms: Operative Management

SUMMARY:
Patients undergoing either operative or non-operative treatment of proximal humerus fractures will be studied with the goal of understanding which treatment modality provides optimal post-injury outcomes.

ELIGIBILITY:
Inclusion Criteria:

* individuals 65 years of age or older with proximal humerus fractures

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (ROM) | at 3 months, 6 months, 12 months, and 24 months from initiation of treatment
  Range of Motion of the shoulder in terms of degrees of motion
  Assessment of forward flexion (0-180 degrees), abduction (0-90 degrees), external rotation (0-90 degrees)
SANE | at 3 months, 6 months, 12 months, and 24 months following initiation of treatment
  "Sane outcome" typically refers to the Single Assessment Numeric Evaluation (SANE) score, a patient-reported outcome measure used in healthcare, particularly in orthopedics. It assesses a patient's perceived function of a joint or body region by asking them to rate it on a scale of 0 to 100, where 100 represents normal function
VAS | at 3 months, 6 months, 12 months, and 24 months following initiation of intervention
  "VAS outcome" refers to the results obtained from using a Visual Analog Scale (VAS). The VAS is a measurement tool, typically a 10 cm or 100 mm line, where individuals indicate the intensity of a subjective experience, such as pain, by marking a point on the line. The distance from one end of the line to the patient's mark is then measured, and this measurement represents the VAS score. A higher score indicates a greater intensity of the experience being measured.
ASES | at 3 months, 6 months, 12 months, and 24 months following initiation of intervention
  The American Shoulder and Elbow Surgeons scale (ASES) is a condition-specific scale that is intended to measure functional limitations and pain of the shoulder. A higher ASES score indicates better shoulder function and less pain, with a score of 100 representing the best possible outcome and a score of 0 representing the worst possible outcome.
EQ-5D-5L | at baseline and subsequently at 3 months, 6 months, 12 months, and 24 months following initiation of intervention
  The EQ-5D-5L score represents a patient's self-reported health status, with values ranging from -0.59 to 1, where 1 indicates the best possible health. It's based on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity. These responses are converted into a single index score using a scoring algorithm.
Brophy/Marx | at baseline and subsequently at 12 months and 24 months after initiation of intervention
  The Brophy-Marx Shoulder Activity Score is a valid and reliable shoulder-specific questionnaire that measures a patient's shoulder activity level over the previous year. The questionnaire generates a numeric score from 0 (least active) to 20 (most active).
PROMIS Social | at 3 months, 12 months, and 24 months following initiation of intervention
  PROMIS, or the Patient-Reported Outcomes Measurement Information System, uses T-scores to represent social health, with a mean of 50 and a standard deviation of 10 for the general US population. Higher T-scores generally indicate a greater amount of the measured concept, such as satisfaction with social roles and activities, while lower scores indicate less.
Radiographic Outcome | at 3 months, 6 months, 12 months, and 24 months following initiation of intervention
  evidence of bony healing, nonunion, or malunion of the fracture on imaging
Complication Rate | at 3 months, 6 months, 12 months, and 24 months following initiation of intervention
  Rate of complications following initiation of management

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Chan, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided